CLINICAL TRIAL: NCT03833037
Title: Observational, Descriptive and Retrospective Study of a Cohort of 90 Consecutive Cases of Synovial Sarcoma Treated in the Orthopedic Surgery Unit of the Orthopedic Surgery and Traumatology Department of the Hospital de Sant Pau Between the Years 1983 and 2016 ( 35 Years)
Brief Title: Study of a Cohort of Cases of Synovial Sarcoma Treated in the Orthopedic Surgery and Traumatology Department of the Hospital de Sant Pau Between 1983 and 2016
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-SAR-2018-100
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Soft Tissue Sarcoma Adult
Keywords: Synovial sarcoma
MeSH Terms: conditions — Sarcoma, Synovial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 23 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Soft tissue sarcomas in adults — Adult sinovial sarcoma

SUMMARY:
The main objectives of this study are the following: to describe the prognostic factors of survival of synovial sarcoma in patients treated by the orthopedic surgery unit oncologic of the orthopedic surgery and traumatology service of the Hospital de Sant Pau during the years 1983-2016.

DETAILED DESCRIPTION:
Another objectives of this Study are:

To analyze exhaustively a series of cases of synovial sarcoma (as an example of classic subtype of soft tissue sarcoma) to analyse the complementary tests performed and their evolution over time.

To analyse the results of surgical treatment and adjuvant therapies in synovial sarcoma and its evolution over time.

To study the prognostic factors dependent on the patient and the applied therapeutics.

To establish a results-based treatment and follow-up algorithm for patients diagnosed with synovial sarcoma.

To describe the epidemiological characteristics of the group of patients in the study.

To evaluate the overall survival and disease-free survival as well as the mortality of the disease.

To assess the rate of local recurrence and remote dissemination of synovial sarcomas in the series.

To demonstrate the influence of neoadjuvant chemotherapy and radiotherapy in the treatment of the tumor.

Conduct a study by age group with respect to the influence on patient survival. To carry out a study by tumor-sized groups with respect to the influence on the survival of the patients.

To carry out a chronological study on the influence of the advances in the treatments on the survival of the patients.

Compare the results obtained with the published literature.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria were: diagnosed cases of synovial sarcoma by the service of pathological anatomy and treated by unit orthopedic surgery oncology, in location of limbs, paravertebral trunk and/or pelvis. We studied the complete medical history of the cases available for the analysis and with a minimum follow-up of 12 months.

Exclusion Criteria:

Ages: 10 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The overall sample size will be 90 cases of synovial sarcoma diagnosed and treated by the unit, considering a sufficient number of cases in the analysis with sufficient potency to respond to the issues raised methodology. Sources of information all clinical records of the patients will be reviewed and a total of 104 elements collected, collecting data in relation to the epidemiology, personal and family history, physical examination, complementary tests of Local and extension diagnosis, time to diagnosis and treatment, pathological diagnosis, surgical technique, adjuvant therapy, complications of treatment, staging, clinical evolution, recurrences and metastases, functional valuation and data of survival and follow-up.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of cases of synovial sarcoma | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Lamas, Study Director — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided